CLINICAL TRIAL: NCT06983470
Title: Predictive Utility and Mechanisms of Sacral Evoked Responses in Sacral Neuromodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Timothy Bruns, Associate Professor of Biomedical Engineering, Medical School, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00222497
Record Dates: First submitted 2025-05-09; First posted 2025-05-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- VMR followed by SER (Experimental): SNM implants will use parameters selected based on visual-motor responses (VMRs) for four weeks followed by parameters selected based on sacral evoked responses (SERs) for four weeks.
  Interventions: Device: SNM based on visual-motor responses (VMRs); Device: SNM based on sacral evoked responses (SERs)
- SER followed by VMR (Experimental): SNM implants will use parameters selected based on sacral evoked responses (SERs) for four weeks followed by parameters selected based on visual-motor responses (VMRs) for four weeks.
  Interventions: Device: SNM based on visual-motor responses (VMRs); Device: SNM based on sacral evoked responses (SERs)

INTERVENTIONS:
Device: SNM based on visual-motor responses (VMRs) — SNM using parameters that elicited the best VMRs in the stage-1 implant procedure
Device: SNM based on sacral evoked responses (SERs) — SNM using parameters that elicited the best SERs in the stage-1 implant procedure

SUMMARY:
Electrical stimulation of the sacral nerve can help with bladder problems and pelvic pain but researchers don't understand exactly how the stimulation helps. The goal of this study is to examine signals evoked during sacral neuromodulation (SNM or electrical stimulation of the sacral nerve) and their relationship to the selection of stimulation parameters that improve pelvic function symptoms. This study uses SNM parameters based on visual-motor responses (VMR) or sacral evoked responses (SER). It is investigating how the parameter selection impacts change in bladder function.

DETAILED DESCRIPTION:
Some surgical procedures will be conducted at the Chealsea Hospital (75 S Main St, Chelsea, MI 48118) and all others will be done at Michigan Medicine facilities.

ELIGIBILITY:
Inclusion Criteria:

* Determined by the research team to be fully eligible to receive a sacral neuromodulation implant at a sacral nerve as part of their normal clinical care for overactive bladder (OAB).
* Adult (18 or older), capable of providing own informed consent and communicating clearly with research team.
* Capable of speaking, reading, and understanding English, as all study questionnaires are standardized assessments only available in English.

Exclusion Criteria:

* Areflexive or atonic bladder.
* Pregnant or planning to become pregnant. If a woman of child-bearing potential wishes to participate in this study, they will be pre-screened with a test to detect pregnancy.
* Diagnosed neurogenic bladder, sacral nerve damage, lower motor dysfunction, or other conditions that would affect the neural circuits involved in micturition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Change in bladder function score during SNM using visual-motor responses (VMR)-selected stimulation programs | Baseline through the conclusion of study participation, approximately 3 months
  Bladder function score is assessed using the American Urological Association Symptom Index. The American Urological Association Symptom Index has a range of 0 (no dysfunction) to 35 (maximum dysfunction). A decrease in score indicates improvement.
Change in bladder function score during SNM using sacral evoked responses (SER)-selected stimulation programs | Baseline through the conclusion of study participation, approximately 3 months
  Bladder function score is assessed using the American Urological Association Symptom Index. The American Urological Association Symptom Index has a range of 0 (no dysfunction) to 35 (maximum dysfunction). A decrease in score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bruns, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No